CLINICAL TRIAL: NCT06962501
Title: The Impact of Acute Oral Ketone Monoester Supplementation on Resting-state Brain Connectivity in Adults With Cognitive Decline
Brief Title: Acute Oral Ketone Monoester Supplementation and Resting-state Brain Connectivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Department of Geriatric Medicine FELIX PLATTER (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Sabine Krumm, PD Sabine Krumm, PhD, University Department of Geriatric Medicine FELIX PLATTER
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02148
Record Dates: First submitted 2025-04-09; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: MCI; SCD
Keywords: keton; MCI; SCD; CBF; DMN

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The impact of acute oral ketone monoester supplementation (Experimental): Single dose of a ketone monoester ([R]-3-hydroxybutyl [R]-3-hydroxybutyrate; 0.3 g β-OHB/kg body weight)
  Interventions: Dietary Supplement: Oral ketone monoester (KME)

INTERVENTIONS:
Dietary Supplement: Oral ketone monoester (KME) — The oral ketone monoester supplement should increase the global CBF and improve resting-state connectivity in the DMN in adults with SCD or MCI. The participants will take one dose of the supplement followed by measurement, to figure out if there are any noticeable changes.

SUMMARY:
The primary objectives of this pilot study are to test if a single dose of an oral ketone monoester supplement will increase blood flow and connectivity in the brain in adults with subjective cognitive decline (SCD) or mild cognitive impairment (MCI).

The main questions it aims to answer are:

Does a single dose of an oral ketone supplement increase global cerebral blood flow (CBF)?

Does a single dose of an oral ketone supplement improve resting-state functional connectivity in the Default Mode Network (DMN)?

Does the increase in CBF positively correlate with improved functional connectivity in the DMN?

Participants will:

* Attend one 2-hour session, which includes:
* Neurocognitive assessment
* MRI Scans (two, each 15 Minutes)
* Capillary blood ketone level measurements
* Hemodynamic assessment (blood pressure, heart rate)

DETAILED DESCRIPTION:
In this non-randomized, single-arm study participants will undergo a baseline MRI scan to assess functional connectivity in the DMN and resting CBF without ketone supplementation. Participants will then consume 0.3 g/kg body weight of a ketone monoester supplement (∆G Tactical) and then rest for 70 minutes. Participants will then undergo a second MRI scan to evaluate changes in functional connectivity and CBF, with capillary β-OHB and blood pressure measured before and after each scan. The entire experimental visit, including scans and assessments, will last up to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 years or older
* Subjective Cognitive Decline (SCD) or Mild Cognitive Impairment (MCI)

SCD CRITERIA:

* Self-experienced, persistent decline of cognitive abilities within the last 5 years in relation to a previously normal status
* Normal results on demographically adjusted standardized cognitive tests
* Accompanied by concerns associated with SCD and a feeling of worse performance than others in the same age group
* Decline must not be related to a specific event or explained by a specific disease, medical disorder, medication, or substance abuse

MCI CRITERIA

* Fulfils criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5):
* Demographically adjusted performance between -1 and -2 SD below average in one or more cognitive domains on standardized cognitive tests
* Accompanied by concern from the individual, a knowledgeable informant, or clinician indicating mild cognitive decline
* Capacity for independent daily activities is maintained

Exclusion Criteria:

* Clinical diagnoses of psychiatric disorders (e.g., anxiety disorders, depression)
* Diagnosed major neurocognitive disorder (i.e., dementia)
* Association of SCD or MCI with delirium
* Diagnosed cardiometabolic disease (Uncontrolled hypertension (systolic blood pressure >160 mm Hg, and/or diastolic blood pressure >100 mm Hg, Type 2 diabetes)
* Substance use disorder
* History of heart attack or stroke requiring hospitalization in the past 3 years
* MRI contraindications, including implanted medical devices
* Experiencing residual fatigue, brain fog, or tiredness post-acute illness (i.e., long-COVID)
* Severe literacy, visual, hearing, and/or speech impairment that would make participation in the study difficult or impossible
* Individuals who are not fluent in Swiss German or German

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity of the DMN | 90 minutes
  Functional connectivity of the default mode network (DMN) is measured via functional MRI. Changes in BOLD signal in each region are determined by independent component analysis and then functional connectivity is measured as a Pearson correlation (r) between the neural regions comprising the DMN and transformed into a z score.

SECONDARY OUTCOMES:
Cerebral blood flow | 90 minutes
  Sum of blood flow in the internal carotid and vertebral arteries via phase contrast MRI in ml/min.

OTHER OUTCOMES:
Plasma β-OHB | 90 minutes
  Plasma β-OHB will be measured (in millimolar, mM) via finger prick at set intervals before and after supplement ingestion using a handheld commercial analyzer (FreeStyle Libre, Abbott).
Arterial blood pressure | 90 minutes
  Automated blood pressure cuff measurement of brachial artery pressure in mmHg.
Heart Rate | 90 minutes
  Automated blood pressure cuff measurement of heart rate in bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Krumm, PD, PhD, Principal Investigator — University Department of Geriatric Medicine FELIX PLATTER
Locations (1):
- University Hospital of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
Trial and participant data will be handled with uttermost discretion and is only accessible to authorised personnel who require the data to fulfil their duties within the scope of the study.